CLINICAL TRIAL: NCT05571670
Title: Bile Acid and Lipid Metabolism in Patients With Drug-induced Acute Insulin Resistance
Brief Title: Bile Acids in Acute Insulin Resistance
Status: Terminated | Type: Observational
Why Stopped: Poor enrollment
Sponsor: Columbia University (Other)
Responsible Party: Principal Investigator, Joshua Cook, Assistant Professor of Medicine at the Columbia University Medical Center, Columbia University
Other Study IDs: AAAU0504
Record Dates: First submitted 2022-10-05; First posted 2022-10-07 (Actual); Last update posted 2025-01-16 (Actual); Status verified 2025-01

CONDITIONS: PI3K Gene Mutation; AKT Gene Mutation; MTOR Gene Mutation; Cancer; Insulin Resistance
Keywords: Insulin resistance; Bile acids; Cardiovascular disease; Dyslipidemia
MeSH Terms: conditions — Neoplasms; Insulin Resistance; Cardiovascular Diseases; Dyslipidemias

STUDY DESIGN:
Observational Model: Case-Only | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Blood samples will be drawn fasting +/- after 2-hour mixed meal tolerance test immediately before and then at 2 and 4 weeks after initiation of PI3K/AKT/mTOR inhibitor treatment. Blood will also be drawn at the end of treatment if treatment concludes within 2 months of starting.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Patients treated with PI3K/AKT/mTOR inhibitors for cancer: Patients with cancer being treated with PI3K/AKT/mTOR inhibitors will be studied prospectively for the impact of treatment on bile acid metabolism as a function of drug-induced acute insulin resistance. Treatments will be selected by patients' treating oncologist based on standard of care.
  Interventions: Drug: Drug-induced acute insulin resistance due to PI3K inhibitor, AKT inhibitor, or mTOR inhibitor

INTERVENTIONS:
Drug: Drug-induced acute insulin resistance due to PI3K inhibitor, AKT inhibitor, or mTOR inhibitor — Participants will be treated with PI3K/AKT/mTOR inhibitors by their treating oncologist based on standard of care. This study will prospectively monitor bile acids and parameters of insulin resistance before and during treatment with these drugs.

SUMMARY:
This is a prospective observational study with a primary goal of monitoring changes in circulating bile acid profiles and parameters of glucose and lipid metabolism prior, during, and after cancer treatment with agents that directly impair insulin action: PI3K inhibitors, AKT inhibitors, and mTOR inhibitors. Patients will not receive any cancer treatment specifically for the purposes of this study. Rather, this study will be based on treatment decisions made independently by participants' oncologists according to standard of care or other clinical trial protocol. This study seeks to enroll at least 25 participants each for PI3K inhibitors, mTOR inhibitors and, once available for open-label treatment, AKT inhibitors.

DETAILED DESCRIPTION:
The primary objective of this study is to determine the effect of drug-induced acute insulin resistance (diaIR) on the ratio of 12α-hydroxylated bile acids (12-HBA) to 12α-hydroxylated bile acids (non-12-HBA) in cancer patients treated with phosphatidylinositol-4,5-bisphosphate kinase (PI3K) inhibitors (PI3Ki), mammalian target of rapamycin (mTOR) inhibitors (mTORi), and AKT inhibitors (AKTi) once possible. Specifically, this study will: (1) verify the induction of diaIR by monitoring changes in fasting ± postprandial blood glucose, insulin/c-peptide, and fructosamine; and (2) assess qualitative and quantitative changes in the circulating bile acid (BA) pool (including bile acid intermediary metabolites) by mass spectrometry in the fasting ± postprandial states prior to and then at 2 and 4 weeks after starting treatment. This study focuses in particular on determining changes in the 12α-hydroxylated bile acids to 12α-hydroxylated bile acids, as well as each of these subclasses and their individual substituents as a proportion of the overall BA pool.

ELIGIBILITY:
Inclusion Criteria:

* Age ≥ 18 years
* Speaks English and/ or Spanish
* Any cancer diagnosis
* Planned for treatment with:

  * PI3K inhibitors

    * Alpelisib
    * Inavolisib
    * Any experimental PI3K inhibitor
  * AKT inhibitors (if these become available for open-label use during the study course)

    * Afuresertib
    * Capivasertib
    * Ipatasertib
    * Miransertib
    * Uposertib
  * mTOR inhibitors

    * Everolimus
    * Sirolimus
    * Temsirolimus
* Signed informed consent

Exclusion Criteria:

* Known dysglycemia
* Known diagnosis of diabetes mellitus
* Treatment with glucose-lowering medications at baseline

  * Insulin
  * Sulfonylureas or meglitinides
  * Metformin >1000mg total daily dose
  * Thiazolidinediones
  * SGLT2 inhibitors
  * GLP-1 receptor agonists
  * DPP4 inhibitors
  * Amylin mimetics
  * Acarbose
* Significant biochemical evidence of liver dysfunction on lab tests within 30 days before starting drug that have not fallen to below the following thresholds prior to starting drug
* Significant functional or anatomical abnormalities of the small intestine
* Use of certain medications at baseline, within 7 days of starting cancer drug
* Allergy to cow dairy or soy (only excludes from MMTT, does not exclude from fasting blood draws)
* Inability to provide informed consent

Ages: 18 Years to 99 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Adult patients of any gender, without pre-existing diabetes, treated with PI3K/AKT/mTOR inhibitors for cancer according to standard of care.
Sampling Method: Non-Probability Sample
Enrollment: 3 (Actual)
Dates: Start 2022-06-10 (Actual); Primary Completion 2022-06-10 (Actual); Study Completion 2022-06-10 (Actual)

PRIMARY OUTCOMES:
Ratio of 12-HBA to non-12-HBA | 1-2 Months
  Insulin resistance is expected to cause a rise in total bile acids, but with 12-alpha-hydroxylated bile acid (12-HBA) species outpacing non-12-alpha-hydroxylated bile acid (non-12-HBA) species, leading to a rise in the 12-HBA:non-12-HBA ratio. This would indicate that insulin resistance per se is sufficient to alter 12-HBA balance, and thus 12-HBA may be a useful therapeutic target for management of the macrovascular complications of insulin resistance. BA profile and levels of BA intermediates 7-HCO and 7,12-diHCO will be measured by LC-MS/MS when fasting +/- after 2-hour mixed meal tolerance test.
Insulin resistance | 1-2 months
  Determine the timing and extent of PI3K/AKT/mTOR inhibitor treatment on parameters of insulin resistance: glucose, insulin, c-peptide, and adiponectin when fasting +/- following 2-hour mixed meal tolerance test

SECONDARY OUTCOMES:
Lipid profile | 1-2 months
  The primary endpoint is the outcome of the secondary objective: namely, evaluation of the effect of PI3Ki/AKTi/mTORi-induced insulin resistance on the lipid profile (total cholesterol, HDL cholesterol, LDL cholesterol, triglycerides, free fatty acids) when fasting +/- after 2-hour mixed meal tolerance test
Surrogate markers of BA signaling | 1-2 months
  Determine the timing and extent of PI3K/AKT/mTOR inhibitor treatment on parameters of bile acid signaling: fibroblast growth factor 19 (FGF-19) and glucagon-like peptide-1 (GLP-1). We expect that a shift in BA pool composition (especially as regards 12-HBA vs non-12-HBA) will impact differentially on FGF-19 and GLP-1 levels.

CONTACTS AND LOCATIONS:
Locations (1):
- Columbia University Medical Center, New York, New York, United States